CLINICAL TRIAL: NCT04206878
Title: Evaluating the Feasibility of Point of Care Birth Testing in Eswatini
Status: Completed | Type: Observational
Sponsor: Elizabeth Glaser Pediatric AIDS Foundation (Other)
Collaborators: UNITAID (Other)
Responsible Party: Sponsor
Other Study IDs: EG0206
Record Dates: First submitted 2019-03-11; First posted 2019-12-20 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: HIV Infections; HIV/AIDS; Pediatric HIV Infection; Transmission, Perinatal Infection; Infant Morbidity; Neonatal Infection
Keywords: HIV; POC; EID; Pediatrics
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HIV-exposed infants (HEI) eligible for birth testing: All HEI live births born at, or presenting to, one of the 3 study sites, within 3 days of birth.
  Interventions: Diagnostic Test: Point-of-care birth test

INTERVENTIONS:
Diagnostic Test: Point-of-care birth test — Collect quantitative data through clinical chart and form abstractions; collect qualitative data through in-depth interviews with caregivers, health workers and policymakers

SUMMARY:
This study aims to assess the feasibility and utility of birth testing using point-of-care (POC) testing in maternity settings in Eswatini.

DETAILED DESCRIPTION:
This UNITAID-funded study aims to assess feasibility and utility of birth testing, [early infant diagnosis for HIV, (EID)], using point-of-care (POC) HIV nucleic acid testing (NAT) at high volume maternity settings. Birth testing is defined as tests within 3 days of life. Outcome measures will include age at testing, turnaround time from testing to caregiver result receipt, HIV positivity rate, and timing of anti-retroviral therapy (ART) initiation for HIV-positive infants. The study will document retention in care for those who tested positive at birth, and the percent of those who tested negative at birth who returned for six week testing. The study will also assess the feasibility and acceptability of POC birth testing using interviews with policymakers, health care workers and caregivers of HIV-exposed infants (HEI).

ELIGIBILITY:
Inclusion Criteria:

* HIV Exposed Infants

  * Must have been newly born at the study sites or presenting in study sites within 3 days after birth
  * Tested for HIV using POC EID platform (mother or caregiver agreed to have infant tested)
* Health Care Workers (HCWs)

  * HCWs who have used POC EID for at least three months, at project sites
  * HCWs that work directly with POC EID services at maternity providing clinical services or operating the platform
  * HCWs who consent to be interviewed
  * HCWs able to speak one of the study languages
* Laboratory Managers and program leads/focal persons:

  * National or regional level manager or head of department whose responsibilities include EID
  * Member of a national technical working group or advisory board member working on EID
  * National level representative from the MOH
  * Laboratory managers in the 3 study sites
  * Participants 18 years and above who consent to be interviewed
* Mothers/caregivers:

  * Mother/caregiver of an HEI who was offered POC EID at birth
  * Provides consent to participate in the study
  * Is 18 years or older, or is less than 18 years old but is legally married (and thus legally emancipated)
  * Speaks one of the study languages

Exclusion Criteria:

* HEIs:

  * HEI tested for HIV using conventional EID at projects sites
  * HEI whose caregivers refuse birth testing
  * HEI where the clinician deems there is a contra-indication for sample collection for birth testing (e.g. severe hemophilia)
* HCWs:

  * HCWs who work within project sites that do not make use of EID (i.e. HCWs who are not involved directly with EID)
  * HCWs working in non-project sites
  * HCWs who are unable to consent or do not speak a study language
* Laboratory Managers and program leads/focal persons:

  * Inability to give consent
  * Inability to speak study language
* Mothers/Caregivers:

  * Not eligible for POC birth testing services
  * Not able to consent
  * Does not speak English or SiSwati

Max Age: 4 Days | Sex: All
Age Groups: Child
Study Population: For quantitative component:
  1. All HEIs newly born at the selected sites or presenting in study sites within 3 days after birth
     For qualitative component:
  2. Health care workers and phlebotomists who are currently employed in study sites who are involved in providing POC EID services
  3. Laboratory managers and program leads/focal persons at the Ministry of Health
  4. Mothers/caregivers of HEI delivered or presenting in study sites within 3 days after birthwho were offered POC HIV EID testing at birth
Sampling Method: Non-Probability Sample
Enrollment: 3316 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-07-03 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Percent of eligible HEI born at or presenting to pilot facilities who receive POC EID testing at birth | 24 months
  Number of eligible HEI born at or presenting to pilot facilities receiving POC EID testing as a proportion of the number of HEI born or presenting to pilot facilities

SECONDARY OUTCOMES:
Percent of tested HEI whose caregivers receive results of the POC EID birth testing | 24 months
  Number of tested HEI whose caregivers receive results of the POC EID birth testing as a proportion of the number of tested HEI
HIV positivity rate among HEI tested at birth | 24 months
  Number of HEI testing HIV positive at birth as a proportion of the number of HEI tested at birth
Number of HIV-infected infants (HII) tested at birth who are started on ART within 2 weeks of the birth test | 24 months
  Number of HII tested at birth started on ART within 2 weeks as a proportion of the number of HII tested at birth
Percent of HEI testing HIV negative at birth who return for testing at 6-8 weeks | 24 months
  Number of HEI testing HIV negative at birth who return for testing at 6-8 weeks as a proportion of the number of HEI testing HIV negative at birth
Percent of HEI who test HIV negative at birth and who test positive at 6-8 weeks | 24 months
  Number of HEI who test HIV negative at birth and who test HIV positive at 6-8 weeks as a proportion of the number of HEI who test HIV negative at birth
Percent of HII testing HIV positive at birth or at 6-8 weeks in care for the first 3 and/or 6 months of life | 24 months
  The number of HII testing HIV positive at birth or at 6-8 weeks in care for the first and/or 6 months of life as a proportion of the number of HII testing HIV positive at birth or at 6-8 week of life

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Cohn, Study Director — Elizabeth Glaser Pediatric AIDS Foundation
Locations (1):
- Mbabane Government Hospital, Hlathikhulu Hospital, and Good Shepherd Hospital, Mbabane, Eswatini

IPD SHARING:
Plan to Share IPD: No